CLINICAL TRIAL: NCT05566535
Title: Changes in Quality of Life (QoL) and Symptoms in Patients With Polycythemia Vera (PV) Receiving Ruxolitinib (Ruxo) in a Routine Clinical Practice
Brief Title: Changes in QoL and Symptoms in Patients With Polycythemia Vera Receiving Ruxo in a Routine Clinical Practice
Acronym: QoL-PV-R
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Multinational Center for Quality of Life Research, Russia (Other)
Responsible Party: Sponsor
Other Study IDs: CINC424BRU04T
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Polycythemia Vera
Keywords: ruxolitinib; quality of life
MeSH Terms: conditions — Polycythemia Vera | interventions — ruxolitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ruxolitinib — Ruxo will be administered to patients with PV in a real-world setting. Treatment with Ruxo is according to local approved label. Ruxo treatment should be administered according to drug official instruction and in compliance with clinical practice at the certain medical center.

SUMMARY:
The purpose of this multicenter observational prospective cohort study is to examine changes in QoL and symptoms in patients with polycythemia vera (PV) during treatment with ruxolitinib (Ruxo), and to evaluate efficacy and safety of Ruxo in a real-world setting

ELIGIBILITY:
Inclusion Criteria:

* Patients who have confirmed diagnosis of PV
* Patients whose age - 18 years and older
* Patients who signed informed consent
* Patients who able to fill out questionnaires

Exclusion Criteria:

* Patients enrolled in clinical trials
* Patients with contraindications to Ruxo in accordance with instruction for use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with PV will be enrolled after being prescribed with Ruxo. The eligibility criteria for this study are broader than those for patients to be treated with Ruxo in randomized clinical trials, so as to be reflective of routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in QoL as per SF-36 questionnaire domains at 3 and 9 months of Ruxo treatment | Baseline, 3 and 9 months of Ruxo treatment
  The difference in QoL means of SF-36 domains at 3 and 9 months as compared to their Baseline will be analyzed

SECONDARY OUTCOMES:
Change From Baseline in MPN10 Total score over time | Baseline, 1, 3, 6, 9 and 12 months of Ruxo treatment
  The difference in MPN10 Total Symptom Score means by MPN10 at different time-points of Ruxo treatment as compared to their Baseline will be analyzed. Also the percentage of patients with the lowest symptom burden, corresponding to MPN10 Total scores of 0 - 7 (quartile 1), at different treatment time-points (Baseline, 1, 3, 6, 9 and 12 months) will be calculated
Change From Baseline in severity of each symptom by MPN10 over time | Baseline, 1, 3, 6, 9 and 12 months of Ruxo treatment
  The difference in MPN10 symptom score means at different time-points of Ruxo treatment as compared to their Baseline will be analyzed
Percentage of patients achieving a ≥ 50% improvement from Baseline in MPN10 Total Symptom Score over time | 1, 3, 6, 9 and 12 months of Ruxo treatment
  The number of patients with MPN10 Total Symptom Score decrease ≥ 50% at 1, 3, 6, 9 and 12 months of Ruxo treatment as compared to its' Baseline will be calculated
Change From Baseline in QoL as per SF-36 questionnaire domains over 12 months of Ruxo treatment | Baseline, 1, 3, 6, 9 and 12 months of Ruxo treatment
  The difference in QoL means of SF-36 domains at different time-points of Ruxo treatment as compared to their Baseline will be analyzed
The percentage of patients who achieved overall clinicohematologic response at 9 months of treatment with Ruxo | 9 months
  Overall clinicohematologic response will be defined as any participant who achieved a complete or partial clinicohematologic response per the National criteria for response in polycythemia vera (2021) and European LeukNet recommendations (2013). A complete response (CR) will be defined as: hematocrit control (<45%) with the absence of phlebotomy eligibility ≥12 weeks, spleen volume reduction at least 35% from baseline, platelet count less than or equal to 400 x 109/L, and white blood cell count less than or equal to 10 x 109/L, and symptom regress during ≥12 weeks as well as histological remission. A Partial Response (PR) will be defined as all the above criteria excluding histological remission
The Percentage of patients who achieved hematocrit (Hct) control at 9 months of treatment with Ruxo | 9 months
  Hematocrit control is Ht <45% with the absence of phlebotomy eligibility beginning at 3 months visit and continuing through 9 months
The percentage of patients with positive changes of wellbeing during Ruxo treatment | 1, 3, 6, 9 and 12 months of Ruxo treatment
  The number of patients who reported improvement as per Patient Global Impression of Changes scale at different time-points of treatment will be analyzed
The percentage of patients satisfied/dissatisfied with Ruxo treatment over time | 1, 3, 6, 9 and 12 months of Ruxo treatment
  The number of patients satisfied/dissatisfied with treatment according to Patient' Treatment Satisfaction Checklist at different time-points of treatment will be analyzed

IPD SHARING:
Plan to Share IPD: No